CLINICAL TRIAL: NCT03515629
Title: A Randomized, Phase 3, Open-Label Study of Combinations of REGN2810 (Anti-PD-1 Antibody), Platinum-based Doublet Chemotherapy, and Ipilimumab (Anti-CTLA-4 Antibody) Versus Pembrolizumab Monotherapy in First-Line Treatment of Patients With Advanced or Metastatic Non-Small Cell Lung Cancer With Tumors Expressing PD-L1 ≥50%
Brief Title: REGN2810 (Anti-PD-1 Antibody), Platinum-based Doublet Chemotherapy, and Ipilimumab (Anti-CTLA-4 Antibody) Versus Pembrolizumab Monotherapy in Patients With Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-16111; 2017-001041-27 (EudraCT Number)
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stage IIIB; Stage IV; Non-squamous NSCLC; Squamous NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab (Active Comparator): Pembrolizumab
  Interventions: Drug: Pembrolizumab
- REGN2810/ipi (Experimental): REGN2810/ipi
  Interventions: Drug: REGN2810/ipi
- REGN2810/chemo/ipi (Experimental): REGN2810/chemo/ipi
  Interventions: Drug: REGN2810/chemo/ipi

INTERVENTIONS:
Drug: REGN2810/ipi — REGN2810 plus ipilimumab
  Other Names: cemiplimab
  Arms: REGN2810/ipi
Drug: REGN2810/chemo/ipi — REGN2810 plus chemotherapy plus Ipilimumab
  Other Names: cemiplimab
  Arms: REGN2810/chemo/ipi
Drug: Pembrolizumab — Reference drug administered IV infusion
  Arms: Pembrolizumab

SUMMARY:
The primary objective of the study is to compare the progression-free survival (PFS) of REGN2810 (cemiplimab) plus ipilimumab combination therapy (hereinafter referred to as REGN2810/ipi) and REGN2810 plus 2 cycles only of platinum-based doublet chemotherapy plus ipilimumab combination therapy (hereinafter referred to as "REGN2810/chemo/ipi") with standard-of-care pembrolizumab monotherapy in the first-line treatment of patients with advanced squamous or non-squamous non-small cell lung cancer (NSCLC) whose tumors express programmed death ligand 1 (PD-L1) in ≥50% of tumor cells. The key secondary objectives of the study are to compare the overall survival (OS) of REGN2810/ipi and REGN2810/chemo/ipi with pembrolizumab monotherapy in the first-line treatment of patients with advanced squamous or non-squamous NSCLC whose tumors express PD-L1 in ≥50% of tumor cells and to compare the overall response rate (ORR) of REGN2810/ipi and REGN2810/chemo/ipi with pembrolizumab monotherapy in the first-line treatment of patients with advanced squamous or non-squamous NSCLC whose tumors express PD-L1 in ≥50% of tumor cells.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with histologically or cytologically documented squamous or non-squamous NSCLC with stage IIIB or stage IV disease, who received no prior systemic treatment for recurrent or metastatic NSCLC
2. Availability of an archival (≤5 months) or on-study obtained formalin-fixed, paraffin-embedded tumor tissue sample which has not previously been irradiated
3. Expression of PD-L1 in ≥50% of tumor cells determined by the commercially available assay performed by the central laboratory
4. At least 1 radiographically measureable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria. Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
6. Anticipated life expectancy of at least 3 months

Key Exclusion Criteria:

1. Patients who have never smoked, defined as smoking ≤100 cigarettes in a lifetime
2. Active or untreated brain metastases or spinal cord compression
3. Patients with tumors tested positive for Epidermal growth factor receptor (EGFR) gene mutations, Anaplastic lymphoma kinase (ALK) gene translocations, or C-ros oncogene receptor tyrosine kinase(ROS1) fusions
4. Encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
5. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis or organizing pneumonia), of active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management, or of pneumonitis within the last 5 years
6. Ongoing or recent evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk of immune-related treatment-emergent adverse events (irTEAEs)
7. Previous treatment with idelalisib at any time (ZYDELIG®)
8. Patients with a condition requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 14 days of randomization

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- Regeneron Research Site, St. Petersburg, Florida, United States
- Regeneron Research Site, Cremona, Italy
- Regeneron Research Site, Vilnius, Lithuania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 centers that randomized 5 participants in the United States, Lithuania, and Italy.
Pre-assignment Details: Due to program de-prioritization, the sponsor decided to cease enrollment at which time only 5 participants were randomized to 2 of 3 treatment arms (i.e., no participants were randomized to receive pembrolizumab).
Groups:
- Pembrolizumab: Due to ceasing enrollment early, no participants were randomized to receive pembrolizumab.
- Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W: Cemiplimab was administered at 350 mg as an intravenous (IV) infusion every 3 weeks (Q3W) for 108 weeks in combination with ipilimumab administered IV over approximately 90 minutes at 50 mg Q6W for up to 4 doses.
- Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W: Cemiplimab was administered at 350 mg as an IV infusion Q3W for 108 weeks in combination with platinum-based doublet chemotherapy administered IV Q3W for 2 cycles and with ipilimumab administered IV over approximately 90 minutes at 50 mg Q6W for up to 4 doses.
Period: Overall Study
Arm/Group | Pembrolizumab | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Started | 0 | 3 | 2
Completed (Completed study) | 0 | 1 | 1
Not Completed | 0 | 2 | 1
Not completed — Death | 0 | 1 | 1
Not completed — Progressive disease | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF), defined as all enrolled participants who received any amount of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (9.29) | 56.5 (4.95) | 59.6 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by a Blinded Independent Review Committee (IRC) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessments
Description: Per protocol, the final analysis of PFS was to be performed after observing 142 PFS events in the pembrolizumab treatment arm. PFS was not assessed due to insufficient data collected.
Time Frame: Up to 32 months
Population: PFS was not assessed due to insufficient data collected.
Arm/Group | Pembrolizumab | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Per protocol, if the final analysis of PFS was statistically significant for both cemiplimab combination therapy versus pembrolizumab treatment, the analysis of OS for cemiplimab combinations-versus-pembrolizumab comparison was to be performed at the time of PFS analysis, 12 months, and 18 months after analysis of PFS using the same method as used in the analysis of PFS.
Time Frame: Up to 32 months
Population: OS was not assessed due to insufficient data collected.
Arm/Group | Pembrolizumab | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Per protocol, the ORR for each cemiplimab combination-versus-pembrolizumab comparison was to be analyzed using the Cochran-Mantel-Haenszel test stratified by histological status (non-squamous versus squamous).
Time Frame: Up to 32 months
Population: ORR was not assessed due to insufficient data collected.
Arm/Group | Pembrolizumab | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs)
Time Frame: Up to 32 months
Population: Safety analysis set (SAF), defined as all enrolled participants who received any amount of study treatment
Measure: Number; unit: Events
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 3 | 2
Events | 68 | 91

5. Secondary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Time Frame: Up to 32 months
Population: Safety analysis set (SAF), defined as all enrolled participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Any Serious TEAEs
Time Frame: Up to 32 months
Population: Safety analysis set (SAF), defined as all enrolled participants who received any amount of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 3 | 2
Participants | 2 | 2

7. Secondary Outcome: Number of Participants With TEAEs Leading to Death
Time Frame: Up to 32 months
Population: Safety analysis set (SAF), defined as all enrolled participants who received any amount of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 3 | 2
Participants | 1 | 0

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Time Frame: Up to 32 months
Population: Safety analysis set (SAF), defined as all enrolled participants who received any amount of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 3 | 2
Participants | 1 | 1

9. Secondary Outcome: Overall Survival (OS) at 12 Months
Description: as for outcome 2
Time Frame: At 12 months
Population: OS was not assessed due to insufficient data collected.
Arm/Group | Pembrolizumab | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Overall Survival (OS) at 18 Months
Description: as for outcome 2
Time Frame: At 18 months
Population: OS was not assessed due to insufficient data collected.
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Quality of Life (Core 30 Questionnaire)
Description: Quality of Life (QoL) as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) four-point scale, with 1 as "not at all" and 4 as "very much." Per protocol, the change in EORTC QLQ-C30 scores from the first assessment to the end of the study were to be summarized descriptively at each post-baseline time point and compared using a mixed effects model, if appropriate.
Time Frame: Up to 32 months
Population: Due to the minimal amount of responses and decrease in number of overall participants analyzed for this outcome measure, results are not reported to protect the confidentiality of the participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 2 | 2
Score on a scale | NA (NA) — Due to the minimal amount of responses and decrease in number of overall participants analyzed for this outcome measure, results are not reported to protect the confidentiality of the participants. | NA (NA) — Due to the minimal amount of responses and decrease in number of overall participants analyzed for this outcome measure, results are not reported to protect the confidentiality of the participants.

12. Secondary Outcome: Quality of Life (Lung Cancer 13 Questionnaire)
Description: QoL as measured by the Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) to assess lung cancer-associated symptoms and treatment-related side effects among lung cancer patients. The scale for EORTC-QLQ-LC13 is 1-4 for most outcome measures of systems, with 1 rated as "not at all" and 4 rated as "very much." Per protocol, the change in EORTC QLQ-LC13 scores from the first assessment to the end of the study were to be summarized descriptively at each post-baseline time point and compared using a mixed effects model, if appropriate.
Time Frame: Up to 32 months
Population: as for outcome 11
Measure: Median (Standard Deviation); unit: Score on a scale
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
Number analyzed (Participants) | 2 | 2
Score on a scale | NA (NA) — Due to the minimal amount of responses and decrease in number of overall participants analyzed for this outcome measure, results are not reported to protect the confidentiality of the participants. | NA (NA) — Due to the minimal amount of responses and decrease in number of overall participants analyzed for this outcome measure, results are not reported to protect the confidentiality of the participants.

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of study (up to 32 months)
Arm/Group | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W (N=3) | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W (N=2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W (N=3) | Cemiplimab 350 mg Q3W + Chemotherapy + Ipilimumab 50 mg Q6W (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 2 (4) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (3) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (4) | 1 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 1 (1)
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03515629/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT03515629/SAP_001.pdf